CLINICAL TRIAL: NCT00050635
Title: STOP Trial - Sandostatin LAR Depot Trial for the Optimum Prevention of Chemotherapy Induced Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSMS995AUS38; STOP Trial
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Neoplasms; Diarrhea
Keywords: chemotherapy induced diarrhea; diarrhea; CTID; colorectal cancer; Sandostatin LAR Depot; Sandostatin; adverse events; side effects
MeSH Terms: conditions — Neoplasms; Diarrhea; Colorectal Neoplasms | interventions — Octreotide

INTERVENTIONS:
Drug: Sandostatin LAR Depot

SUMMARY:
Currently there is an ongoing clinical trial for patients with chemotherapy induced diarrhea. This trial is being conducted to evaluate the efficacy of two dose levels (30 mg and 40 mg) of an investigational drug in reducing the occurrence of severe (Grade 3 or 4) diarrhea during chemotherapy. Eligible patients must either have experienced NCI Common Toxicity Grade 1 - 4 chemotherapy-induced diarrhea during previous chemotherapy treatment or be experiencing Grade 1-4 chemotherapy-induced diarrhea currently.

In order to participate in this clinical trial, patients must be male or female 18 years of age or older. Inclusion into this investigational drug trial is based on the protocol entry criteria and a detailed evaluation from a participating trial investigator

ELIGIBILITY:
Key Inclusion criteria:

* male or female patients of 18 years of age or older, scheduled or expected to receive at least two cycles of chemotherapy over at least a two- month period as primary or adjuvant therapy for any malignancy,
* have experienced NCI Common Toxicity Grade 1 - 4 diarrhea during previous chemotherapy treatment or are currently experiencing Grade 1-4 diarrhea due to chemotherapy treatment

Key Exclusion criteria:

* females who are pregnant or lactating,
* current use of anticoagulants, except for those who are receiving 1 mg/per day of Coumadin for port maintenance,
* known hypersensitivity to Sandostatin, Sandostatin LAR ® Depot or other related drug or compound,
* history or presence of Crohn™s disease, ulcerative colitis, sprue, or known C. difficile infection, or any other diarrheal syndrome,
* WBC < 3000 /L, Platelets < 75,000 /L, serum creatinine >2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-12; Study Completion 2003-07

PRIMARY OUTCOMES:
Change from baseline and at 6 months in the proportion of patients with NCI Grades 3 and/or 4 diarrhea during chemotherapy

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Kenmar Research Institute, Burbank, California
  - Bay Area Cancer Research Group, Concord, California
  - Compassionate Cancer Care medical Group, Inc., Fountain Valley, California
  - California Cancer Care, Inc., Greenbrae, California
  - Pacific Shores Medical Center, Long Beach, California
  - Kenmar Research Institute, Los Angeles, California
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Pasco Hernando Oncology Associates, New Port Richey, Florida
  - Mid-Florida Hematology & Oncology Centers, PA, Orange City, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - Creticos Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Cancer Care Center, Bloomington, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Delta Oncology, Greenwood, Mississippi
  - Missouri Cancer Associates, Columbia, Missouri
  - Heartland Hematology Oncology Associates, Kansas City, Missouri
  - Arch Medical Services/The Center for Cancer Care and Research, St Louis, Missouri
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - North Shore Hematology Oncology, East Setauket, New York
  - Raleigh Hematology Oncology Associates, Wake Practice, Raleigh, North Carolina
  - Dakota Clinic/Odyssey Research Services, Fargo, North Dakota
  - Nashat Y. Gabrail, MD, Canton, Ohio
  - North Coast Cancer Care, Inc., Sandusky, Ohio
  - Lawrence M. Stallings, MD, Wooster, Ohio
  - Consultants in Medical Oncology-Hematology, Drexel Hill, Pennsylvania
  - Regional Hematology Oncology Assoc, Langhorne, Pennsylvania
  - Oncology Services of Aberdeen, Borden, South Dakota
  - Jones Oncolgy/Hematology Clinic, Germantown, Tennessee
  - McFaddin Ward Cancer - TOPA, Beaumont, Texas
  - Scott & White Hospital/CCPC, Waco, Texas
  - Oncology & Hematology Associates of SW VA, Roanoke, Virginia